CLINICAL TRIAL: NCT02456610
Title: Adoptive Transfer of Peptide Stimulated CMV/EBV Specific Cytotoxic T Lymphocytes to Prevent and Treat EBV/CMV Infections in Patients Post Allogeneic Stem Cell Transplantation in China
Brief Title: Administration of Virus Specific CTLs for the Prophylaxis and Treatment of EBV/CMV Infections After HSCT in China
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-CMV/EBV-CTL
Record Dates: First submitted 2015-05-21; First posted 2015-05-28 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Viral Infection
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infusion of CMV/EBV specific CTLs (Experimental): Repetitive CTLs infusion to treat CMV/EBV activation and infection
  Interventions: Biological: CMV/EBV specific CTLs

INTERVENTIONS:
Biological: CMV/EBV specific CTLs — Patients will receive approximately 1x10e6 CTLs/kg as a single infusion via IV injection and may receive 1 to 8 additional infusions at intervals of one week.

SUMMARY:
Cytomegalovirus (CMV) and Epstein Barr Virus (EBV) cause significant morbidity and mortality in hematopoietic stem cell transplantation (HSCT) patients in China. Antiviral drugs given either prophylactically or as early therapy for patients with detectable viral loads appear to be an effective strategy for reducing viral infections. However, long-term treatment with these drugs is associated with significant toxicity, expense and the appearance of drug resistant virus isolates ultimately resulting in treatment failure. CMV and EBV specific T cells infusion to immunocompromised patients following HSCT is able to induce a successful anti-viral response. The primary purpose of this study is to determine the safety and efficacy of the infusion of CMV and EBV specific cytotoxic T cells (CTLs) for patients with CMV and EBV reactivation or infection.

DETAILED DESCRIPTION:
To generate CMV/EBV specific CTLs, G-CSF mobilized hemopoietic progenitor cell (G-HPC) products or nonmobilized peripheral blood apheresis collectings were stimulated with CMV/EBV specific peptides covering most HLA alleles among Chinese populations. Once the investigators made sufficient numbers of T cells, they tested their ex vivo properties.Then a fraction of CTLs were separated for immediate infusion and the others were frozen for further infusion.

If the donor was available, the donor derived CTLs were started to produce when CMV reactivation was detected by qPCR in recipients peripheral blood. Otherwise, autologous CTLs were used. For patients at high risk of developing CMV/EBV infections after stem cell transplantation, a small part of G-HPC products was extracted for CTLs generation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any type of allogeneic HSCT
* CMV, adenovirus or EBV activation or infection which is defined as below. EBV/CMV reactivation is defined as CMV/EBV DNA levels > 1000 IU/ml for a single test or > 500 IU/ml for two consecutive tests. EBV/CMV related disease were defined as the demonstration of CMV/EBV biopsy specimen or clinical diagnosis through symptoms, signs or radiography.
* Written informed consent and/or signed assent line from patient, parent or guardian
* Positive CMV or EBV serology of the donor
* Absence of severe renal disease (Creatinine > 3x upper limit normal)
* Absence of severe hepatic disease (Bilirubin > 3x upper limit normal, AST > 3x upper limit normal)
* Life expectancy > 30 days

Exclusion Criteria:

* Active acute GVHD grades II-IV
* Received donor lymphocytes infusion(DLI) within 30 days
* Received ATG or other immunosuppressive monoclonal antibodies within 30 days
* Uncontrolled acute infections
* Active and relapse of malignancy
* Received steroids treatment more than 0.5 mg/kg/day prednisone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Toxicity of adoptive transfer of CMV/EBV specific CTLs(The increase of temperature by 1℃ and/or the appearance of rash within 24h after infusion) | 24 hours
  Assessment of acute transfusion toxicity within 24 hours after adoptive CTLs transfer
Assessment of viral load response to the CTL infusion assessed by CMV/EBV specific PCR of peripheral blood | 3 months
  Assess the effect of the CTL infusion on viral load

SECONDARY OUTCOMES:
The incidence of Ⅱ~Ⅳ°aGVHD within 30 days after the last dose of CTL infusion | 3 months
Reconstitution of antiviral immunity monitored by flow cytometry | 6 months
Number of patients with chronic GVHD | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chen Hu, M.D., Ph.D., Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, Beijing Municipality, China